CLINICAL TRIAL: NCT00375752
Title: Neoadjuvant Therapy for Postmenopausal Women With ER and/or PgR Positive Breast Cancer. A Randomized Open Phase II Trial Evaluating the Efficacy of a 6 Months Preoperative Treatment With Letrozole (2.5 mg/Day) With or Without Zoledronic Acid (4 mg Every 4 Weeks)
Brief Title: Efficacy and Safety of Letrozole vs. Letrozole Plus Zoledronic Acid as Endocrine Therapy Before Surgery in Postmenopausal Patients With Breast Cancer
Acronym: FEMZONE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446GDE19; 2004-004007-37 (EudraCT Number)
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; Anti tumor potential; Letrozole; Zoledronic acid; Neoadjuvant treatment; Hormone responsive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open-label, multicenter, randomized
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole (Active Comparator): Letrozole 2.5 mg/day oral letrozole for approximately 6.5 months neoadjuvent treatment
  Interventions: Drug: Letrozole
- Zolendronic Acid + Letrozole (Experimental): 2.5 mg/day oral letrozole for approximately 6.5 months neoadjuvant treatment plus zoledronic acid 4 mg i.v. q4w
  Interventions: Drug: Letrozole; Drug: Zolendronic Acid

INTERVENTIONS:
Drug: Letrozole — 2.5 mg.tablet.
Drug: Zolendronic Acid — 4 mg or an adjusted dose based on renal function in 100 ml physiologic (o.9%) normal saline, (as an intravenous infusion over no less than 15 minutes)
  Arms: Zolendronic Acid + Letrozole

SUMMARY:
This study will evaluate the safety/efficacy of zoledronic acid when given by intravenous infusion every 4 weeks in addition to letrozole as endocrine therapy in postmenopausal patients with hormone responsive breast cancer

DETAILED DESCRIPTION:
Open-label, multicenter, randomized phase II trial over approx 6.5 months of neoadjuvant treatment with letrozole with or without zoledronic acid in postmenopausal patients with primary breast cancer. A total of approximately 850 patients were originally planned to be enrolled; primary study endpoint was the objective response rate (according to modified RECIST criteria) after 6 months of treatment. After the core study, patients willing to participate were followed-up for further 5 years.

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal women with primary invasive breast cancer, histologically confirmed by core needle biopsy, whose tumors are estrogen (ER) and / or progesterone (PgR) positive
* Clinical Stage T1c (Size ≥ 1.5 cm), T2, T3, T4a, b, c, N0 or N1, M0 (TNM Classification). According to the modified RECIST criteria, tumors of size ≥ 1.5 cm are considered measurable by mammography and can be determined as target lesions).
* Tumor measurable by mammography, sonography and clinical examination.
* Adequate bone marrow, renal and hepatic function
* Good health status (ECOG Performance status of 0, 1 or 2)

Exclusion criteria:

* Prior treatment with letrozole or bisphosphonates. Prior and concomitant anti-breast-cancer treatments such as chemotherapy, immunotherapy / biological response modifiers (BRM's), endocrine therapy other than letrozole (including steroids), and radiotherapy. Patients who have received hormone replacement therapy (HRT) will NOT be excluded, provided that HRT is discontinued at least 2 weeks prior to entry into the study.
* Patients with unstable angina, or uncontrolled cardiac disease (e.g. Class III and IV New York Heart Association's Functional Classification, see Appendix 9) or uncontrolled endocrine disorders.
* Evidence of inflammatory breast cancer or distant metastasis.
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures. Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants).
* History of diseases with influence on bone metabolism, such as Paget's disease, Osteogenesis Imperfecta, and primary or secondary hyperthyroidism within the 12 months prior to study entry

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2010-12-16 (Actual); Study Completion 2010-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (23):
- Germany (23):
  - Novartis Investigative Site, Amberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Böblingen
  - Novartis Investigative Site, Celle
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Ebersberg
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamelin
  - Novartis Investigative Site, Hanau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Kempten
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Rheinfelden
  - Novartis Investigative Site, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole (LET): Letrozole 2.5 mg/day oral letrozole for approximately 6.5 months neoadjuvent treatment.
- Letrozole +Zoledronic Acid (LET+ZOL): 2.5 mg/day oral letrozole for approximately 6.5 months neoadjuvant treatment plus zoledronic acid 4 mg i.v. q4w
Period: Overall Study
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL)
Started | 79 | 89
Completed | 67 | 74
Not Completed | 12 | 15
Not completed — Lack of Efficacy | 4 | 4
Not completed — Adverse Event | 1 | 6
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Abnormal Laboratory Value(s) | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Administrative Problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL) | Total
Number analyzed (Participants) | 79 | 89 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (8.4) | 71.3 (9.2) | 70.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 89 | 168
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate (Complete Response (CR) or Partial Response (PR)) Based on MRI- or Mammography and/or Sonography According to Modified RECIST Criteria at Month 6
Description: Sum of longest diameter for all target lesions was reported as baseline sum LD. Baseline sum LD was used as reference to characterize objective tumor response. Response Evaluation Criteria in Solid Tumors has 4 response categories. CR (complete response) = disappearance of all target lesions, PR (partial response)= 30% decrease in sum of longest diameter of target lesions, PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions and SD(stable disease)=small changes that do not meet criteria. Analysis was underpowered due to insufficient recruitment rate.
Time Frame: 6 months
Population: The modified intent-to-treat (mITT) population included all patients of the ITT population for whom at least one post-baseline assessment of tumor response according to modified RECIST made by central review was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL)
Number analyzed (Participants) | 66 | 65
percentage of participants | 54.5 [41.8 to 66.9] | 69.2 [56.6 to 80.1]
Statistical Analysis 1: Comparison: Letrozole (LET) vs Letrozole +Zoledronic Acid (LET+ZOL); Test type: Superiority or Other; p = 0.106, Fisher Exact; Odds Ratio (OR) = 14.7, 95% CI 2-sided [-1.8 to 31.1]

2. Secondary Outcome: Best RECIST Response Based on Central Review at 6 Mos
Description: Best response is defined as the best response the patients has reached during the 6 months of treatment. Response Evaluation Criteria in Solid Tumors (RECIST) has 4 response categories. CR (complete response) = disappearance of all target lesions, PR (partial response) = 30% decrease in the sum of the longest diameter of target lesions, PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions and SD (stable disease) = small changes that do not meet criteria.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL)
Number analyzed (Participants) | 66 | 65
Participants
  Complete Response (CR) | 0 | 2
  at least Paratial Response (PR) | 36 | 43
  at least Stable Disease (SD) | 30 | 19
  Progressive Disease | 0 | 1

3. Secondary Outcome: Number of Patients With Breast Conserving Surgery at 6 Months
Time Frame: Every 6 months
Population: The intent-to-treat (ITT) population included all patients of the safety population for whom at least one post-baseline assessment of tumor response according to the modified RECIST (local or central assessment) was available. During different time points, participants with observations at that timepoint were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL)
Number analyzed (Participants) | 75 | 81
Participants
  Surgery performed | 66 | 77
  Radical mastectomy | 10 | 12
  Modfied radical mastectomy | 3 | 8
  Lumpectomy/Quadrantectomy | 50 | 56
  Lumpectomy/Quadrantectomy + Other | 1 | 1
  Other | 2 | 0

4. Secondary Outcome: Change From Baseline in Tumor Size (Longest Diameter) at Month 6
Description: Tumor size (sum of longest diameter)was analyzed based on the diameters values provided with the central review.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL)
Number analyzed (Participants) | 66 | 65
cm | -1.12 (0.92) | -1.37 (0.96)

5. Secondary Outcome: Mean Changes From Baseline in FACT-B Total Score at 6 Months (ITT, Data as Observed)
Description: The FACT-B total score is calculated by summing all five unweighted subscale scores, with total scores in the range of 0-144.To Derive a FACT-B total score: all sections added together The higher the score the better the QoL
  * + __________ + __________ + __________ + __________ =________=FACT-B Total score (PWB score) (SWB score) (EWB score) (FWB score) (BCS score)
Time Frame: baseline and 6 mos
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Letrozole (LET) | Letrozole +Zoledronic Acid (LET+ZOL)
Number analyzed (Participants) | 67 | 68
score on a scale
  Baseline | 113.3 (16.6) | 109.5 (20.2)
  Month 6: number analyzed (Participants) | 64 | 58
  Month 6 | 112.0 (19.6) | 108.2 (20.5)

ADVERSE EVENTS:
Time Frame: through study completion
Groups:
- Letrozole Plus Zoledronic Acid: 2.5 mg/day oral letrozole for approximately 6.5 months neoadjuvant treatment plus zoledronic acid 4 mg i.v. q4w
Arm/Group | Letrozole | Letrozole Plus Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 3/79 | 14/89
Other Adverse Events (participants affected / at risk) | 56/79 | 67/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=79) | Letrozole Plus Zoledronic Acid (N=89)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 3
Performance status decreased (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=79) | Letrozole Plus Zoledronic Acid (N=89)
Vertigo (Ear and labyrinth disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 10
Dry mouth (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 8 | 12
Chills (General disorders) | 0 | 5
Fatigue (General disorders) | 13 | 20
Pyrexia (General disorders) | 1 | 5
Nasopharyngitis (Infections and infestations) | 7 | 4
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Headache (Nervous system disorders) | 8 | 8
Depression (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 3 | 6
Sleep disorder (Psychiatric disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Hot flush (Vascular disorders) | 25 | 19

LIMITATIONS AND CAVEATS:
Study terminated after 178 patients screened and 168 randomized, due to insufficient recruitment rate (no safety issues decided the reason to terminate study). LPLV for study was on 13-DEC-2010. LPLV of the 5-year follow-up period was on 03-FEB-2016.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e.,data from all sites)in the clinical trial.